CLINICAL TRIAL: NCT05870566
Title: UV Light-mediated Corneal Crosslinking as (Lymph)Angioregressive Pretreatment to Promote Graft Survival After Subsequent High-risk Corneal Transplantation [CrossCornealVision]
Brief Title: Pretreatment to Promote Graft Survival After Subsequent High-risk Corneal Transplantation [CrossCornealVision]
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claus Cursiefen (Other)
Collaborators: Uniklinik Köln, Zentrum für Klinische Studien (Unknown); Uniklinik Köln, Institut für Medizinische Statistik und Bioinformatik (Unknown); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Claus Cursiefen, Prof. Dr., University of Cologne
Organization: University of Cologne (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-5045; 01KG2127 (Other Grant/Funding Number: German Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Corneal Transplantation
Keywords: Cornea; Transplantation; Prevascularized Corneas; Corneal crosslinking with UV light irradiation
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open randomized parallel-group trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal Crosslinking (CXL) (Experimental): In the intervention group, the study intervention (CXL) will be administered to stabilize therecipient cornea (which remains in place after penetrating keratoplasty) and to reduce CoNV 8 to 10 weeks prior to corneal transplantation. The study intervention will be repeated once (after 4 weeks prior to transplantation at the latest at the earliest) if insufficient (less than 50%) reduction of CoNV should be observed (to be decided by the respective surgeon). (Protocol V04_0 Page 45) Corneal transplantation will be performed as standard full-thickness penetrating procedure, and the graft (6.5 to 8.25 in diameter) will be secured with 16-24 interrupted single or 2 double running 10-0 nylon sutures (decision by the surgeon). In case of residual CoNV in the intervention group, visible vessels will may be thermally occluded by fine needle diathermy to avoid intraoperative bleeding and reduce complications (to be decided by the respective surgeon at start of surgery). (Protocol V04_0 Page 46)
  Interventions: Device: Corneal Crosslinking
- control group (No Intervention): In the control group subjects will be directly scheduled for corneal transplantation without previous CXL. A sham CXL procedure will not be performed. Corneal transplantation will be performed as standard full-thickness penetrating procedure, and the graft (6.5 to 8.25 in diameter) will be secured with 16-24 interrupted single or 2 double running 10-0 nylon sutures (decision by the surgeon). In case of residual CoNV in the intervention group, visible vessels will may be thermally occluded by fine needle diathermy to avoid intraoperative bleeding and reduce complications (to be decided by the respective surgeon at start of surgery). In the control group, no fine needle diathermy will be performed, as this procedure combined with corneal transplantation in previously non-crosslinked eyes might lead to fistulas and thereby to potential intraocular infections. (Protocol V04_0 Page 46)

INTERVENTIONS:
Device: Corneal Crosslinking — Riboflavin isotonic, 0,1 % Vitamin B2, with Dextran 20,0%, for epi-off procedure or Riboflavin isotonic 0,1% (Vitamin B2), 1,1% HPMC without Dextran for epi-off) 0.1% riboflavin-5-phosphate and 20% dextran T-500) will be applied to the cornea after epithelial debridement every 2 min for 10 minutes before irradiation and every 2 minutes during the course of a 10 minute exposure to 365 nm UV-A with an irradiance rate of 9 mW/cm2. This dose, mode and scheme of the intervention follows the internationally recognized "accelerated CXL protocol" (Elbaz et al. 2014). The data existing shows equivalent outcome regarding efficacy and safety compared to the standard protocol. To avoid any damage to the limbal stem cells, the limbus will not be irradiated during the procedure, as a CXL device (with maximal diameter of 11 mm) will be used. Furthermore, the limbal area will additionally be protected by a custom-cut LSC protection shield. (Protocol V04_0 Page 45-46)
  Arms: Corneal Crosslinking (CXL)

SUMMARY:
The trial evaluates the effect of corneal crosslinking as pre-treatment before corneal transplantation. The goal is to improve graft survival by reducing pathological vessels through pre-treatment.

DETAILED DESCRIPTION:
Multicenter, two armed, controlled, open randomised parallel-group study to evaluate the effect of corneal crosslinking as pre-treatment vs. no pre-treatment ahead of full-thickness penetrating corneal transplantation.

After screening of inclusion and exclusion criteria, eligible subjects will be included after obtaining informed consent. Randomisation will be performed at a 5:4 ratio. (Protocol V04_0 Page 37) At the baseline assessment, a slit lamp examination and photo documentation as well as LaserFlareCellMeter (if available), corneal tomography, and Slit lamp Adapted Optical Coherence Tomography (SL-OCT) measurements will be performed. In addition, visual acuity and a vision-related quality of life will be assessed. Concomitant medication will be documented. Macula OCT will be performed if deemed necessary. In the intervention arm, the study intervention (CXL) will then be administered to reduce CoNV 10-8 weeks prior to corneal transplantation. Two weeks after CXL a control will be performed including AE documentation, slit lamp examination, SL-OCT, corneal tomography, visual acuity and photo documentation. The study intervention will be repeated once if insufficient (less than 50%) reduction of CoNV should be observed (4 weeks prior to corneal transplantation at the latest). All subjects in the intervention arm will then undergo for corneal transplantation. In the control arm, subjects will be directly scheduled for corneal transplantation. Corneal transplantation will be performed as standard full-thickness penetrating procedure, and the graft (6.5 - 8.25 mm 7.75 mm in diameter) will be secured with 16-24 interrupted single or double running 10-0 nylon single sutures (decision by the surgeon). Postoperatively, follow-up assessments will be performed at 3, 6, 12, 18, and 24 months for all subjects (postoperative visits at these time points are standard of care). A slit lamp examination, concomitant medication, AE and photo documentation as well as LaserFlareCellMeter (if available), corneal tomography, SL-OCT, and corneal endothelial cell count measurements will be performed. In addition, visual acuity and a vision-related quality of life will be assessed. Macula OCT will be performed if deemed necessary. If a subject has any complaints, he or she can contact the responsible trial site at any time.

After consultation with the investigator, additional visits can be scheduled. (Protocol V04_0 Page 50)

ELIGIBILITY:
Inclusion Criteria:

Medical condition or disease to be investigated:

- Pathologically prevascularized cornea with need for corneal transplantation

Further inclusion criteria:

* Written informed consent by subject and/or witness prior to any study-related procedures
* Adult male and female subjects ≥ 18 years old
* ≥ 2 corneal quadrants covered by pathological corneal neovascularization
* Absence of other clinical contraindications to any part or product of the treatment plan
* A cooperative attitude to follow up the study procedures
* In case of bilateral disease only one eye will be included
* Steroid responders with adequate control regiment or local/systemic therapy can be included

Exclusion Criteria:

* < 2 corneal quadrants covered by pathological neovascularization
* Corneal stromal thickness below 400 μm (except in the central 8 mm zone which will be replaced later by a new corneal transplant with new endothelium); peripheral stromal thinning below 400 μm in weakened recipient areas is acceptable for CXL if not affecting more than 50% of the corneal circumference (allowing for later endothelial repopulation)
* Active or suspected intraocular inflammation
* Active corneal ulceration
* Compromised eyelid mobility and/or symblepharon
* Allergy, sensitivity or intolerance to riboflavin or UV
* Contraindications, other than steroid response to the local or systemic antibiotics and/or corticosteroids (other than steroid response) foreseen by the protocol
* Contraindications to the surgical protocol
* Clinically significant or unstable concurrent disease or other medical condition affecting grafting procedure
* Rheumatic diseases treated with systemic immunosuppressive medication
* Subjects unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments
* Participation in another clinical trial where an investigational drug was received less than 4 weeks prior to screening visit
* Positive for human immunodeficiency virus (HIV)
* Known abuse of alcohol, drugs, or medicinal products
* Evidence of any other medical conditions (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the subject's compliance, or place the subject at high risk of complications related to the treatment
* Employees of the sponsor, or employees or relatives of the investigator.
* Pregnant women and nursing mothers as corneal transplantation in standard care is performed under general anaesthesia
* Persons held in an institution by legal or official order
* Dysregulated glaucoma with IOP > 25 mmHg at baseline despite local therapy

(Protocol V04_0 Page 43)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
First episode of endothelial graft rejection | within 24 months after transplantation
  Endothelial graft rejection episode is defined by at least 2 of the following criteria: new endothelial precipitates, new anterior chamber cells/flare, new focal or diffuse edema of the graft. All signs will be analyzed by slit lamp examination, on standardized digital slit lamp pictures, by LaserFlareCellMeter (if available), SL-OCT and corneal tomography. (Protocol V04_0 Page 48)

SECONDARY OUTCOMES:
Regression of CoNV | prior to and 2-4 weeks after each CXL, prior to transplantation and at 3, 6, 12, 18 and 24 months
  Assessed by morphometrical analysis of the corneal area covered by CoNV prior to and 2-4 weeks after each CXL, prior to transplantation and at 3, 6, 12, 18 and 24 months using digital standardized slit lamp images and an independent reading center (CORIC). Note: the corneal area covered by CoNV will also be measured in control patients (not receiving angioregressive CXL) at all visits to determine the natural course of CoNV. (Protocol V04_0 Page 48)
Regression of CoNV | before transplantation
  Number of CXL procedures needed for >50% regression of CoNV
Recurrence of CoNV | after CXL and 3, 6, 12, 18 and 24 months after transplantation
  After CXL and after transplantation
Overall functional graft survival rate | 3, 6, 12, 18 and 24 months after transplantation
  Functional survival of graft will be assessed at every follow-up visit after transplantation clinically and using digital slit lamp pictures, SL-OCT and corneal tomography (for graft thickness) as well as endothelial cell counts
Absence of rejection-related graft failure | 3, 6, 12, 18 and 24 months after transplantation
  Rejection-related graft failure assessed at every follow-up visit after transplantation and defined according to the respective criteria for graft rejection and associated graft failure
Best corrected visual acuity (BCVA) | Prior to CXL, prior to transplantation and after 3, 6, 12, 18, and 24 months
  Best corrected visual acuity (BCVA) in the study eye and BCVA or spectacle corrected visual acuity in the partner eye: assessed at the following time-points: prior to CXL, at control visit after CXL, prior to transplantation and after 3, 6, 12, 18, and 24 months using ETDRS charts (logMAR transformed).
Vision-related quality of life | Prior to CXL, prior to transplantation and after 3, 6, 12, 18, and 24 months
  Overall composite score measured using the NEI-VFQ25 at the following time-points
Active infectious keratitis or corneal ulceration | every study visit
  Clinical assessment by slit lamp examination
Graft dehiscence | 3, 6, 12, 18 and 24 months after transplantation
  Graft dehiscence with leakage of aqueous humor from the graft/host interface, assessed by slit lamp examination
Delayed epithelial wound healing | 3, 6, 12, 18 and 24 months after transplantation
  assessed by slit lamp examination

CONTACTS AND LOCATIONS:
Overall Officials: Claus Cursiefen, Prof. Dr., Principal Investigator — University Hospital of Cologne, Centre for Ophthalmology
Locations (7):
- Germany (7):
  - Augenklinik des Klinikums der Universität München, München, Bavaria
  - University Hospital of Cologne, Centre for Ophthalmology, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Klinik für Augenheilkunde, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Klinik für Augenheilkunde, Homburg, Saarland
  - Charité - Universitätsmedizin Berlin, Klinik für Augenheilkunde, Berlin
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Klinik und Poliklinik für Augenheilkunde - Universitätsmedizin Rostock, Rostock

REFERENCES:
- [Derived] Wiedemann J, Hos D, Limburg E, Zettelmeyer U, Schiller P, Franklin J, Bachmann B, Bohringer D, Dietrich-Ntoukas T, Fuchsluger TA, Geerling G, Lang SJ, Mayer WJ, Priglinger S, Reinhard T, Seitz B, Cursiefen C. UV light-mediated corneal crosslinking as (lymph)angioregressive pretreatment to promote graft survival after subsequent high-risk corneal transplantation (CrossCornealVision): protocol for a multicenter, randomized controlled trial. Trials. 2024 Mar 6;25(1):169. doi: 10.1186/s13063-024-08011-1. PMID 38448965